CLINICAL TRIAL: NCT03972358
Title: Assessing Acceptability and Use of Medical Menstrual Regulation in the United States
Brief Title: Assessing Medical Menstrual Regulation in the United States
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gynuity Health Projects (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 8002
Record Dates: First submitted 2019-05-28; First posted 2019-06-03 (Actual); Last update posted 2021-03-24 (Actual); Status verified 2021-03

CONDITIONS: Menstrual Regulation
MeSH Terms: interventions — Mifepristone; Misoprostol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Medical menstrual regulation (Experimental): Mifepristone 200 mg orally on day 1.
  Misoprostol 800 mcg buccally on day 2 (24 hours after mifepristone).
  Interventions: Drug: Mifepristone; Drug: Misoprostol

INTERVENTIONS:
Drug: Mifepristone — All participants will receive 200 mg mifepristone, to be taken orally on day 1.
Drug: Misoprostol — All participants will receive 800 mcg misoprostol, to be taken buccally 24 hours after mifepristone (day 2)

SUMMARY:
This study will assess the acceptability and use of medical menstrual regulation among women in the United States.

DETAILED DESCRIPTION:
Medical menstrual regulation (MMR) entails the use of uterine evacuation medications by women with late menses without confirming pregnancy status. Provision of MMR in the United States could expand reproductive choice and service options for women. This study will collect data on the acceptability, efficacy, safety and feasibility of MMR among women with missed menses of 1-21 days

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-49 years
2. General good health
3. Does not want to be pregnant
4. Does not want to verify pregnancy status at the study site
5. History of regular monthly menstrual cycles
6. Missed menses of 1-21 days
7. Sexual activity in the past 2 months
8. Willing and able to sign consent forms
9. Willing to provide urine sample at enrollment
10. Willing to return for a follow-up visit

Exclusion Criteria:

1. Known allergies or contraindications to mifepristone and/or misoprostol
2. Symptoms of or risk factors for ectopic pregnancy
3. Current use of an IUD, contraceptive implant or injectable

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 284 (Estimated)
Dates: Start 2020-02-12 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants who report that MMR was acceptable or highly acceptable during the exit interview | Up to 28 days after mifepristone administration
  Acceptability of MMR

SECONDARY OUTCOMES:
Number of participants not pregnant at follow-up | Up to 28 days after mifepristone administration
  Efficacy
Number of participants with adverse events and/or side effects | Up to 28 days after mifepristone administration
  Safety and side effects
Perceived advantages and disadvantages of MMR as reported by participants during the exit interview | Up to 28 days after mifepristone administration
  Experiences, perceived advantages and disadvantages

CONTACTS AND LOCATIONS:
Overall Officials: Wendy R Sheldon, PhD, Principal Investigator — Gynuity Health Projects
Locations (2):
- United States (2):
  - Carafem Health Center, Skokie, Illinois
  - Carafem Health Center, Chevy Chase, Maryland

IPD SHARING:
Plan to Share IPD: No
Sharing de-identified data will be considered upon individual request.